CLINICAL TRIAL: NCT00789516
Title: The Change of Coagulation Markers in Children With β-thalassemia Disease After Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nongnuch Sirachainan, Associate Prof, Mahidol University
Other Study IDs: ID11-48-16
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Thalassemia
Keywords: Coagulation markers, thalassemia disease post SCT
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Normal control
- 2: B thalassemia regular transfusion
- 3: B thalassemia post transplantation

SUMMARY:
Hypercoagulable state is well recognized in patients with β-thalassemia. Evidences of hypercoagulability include abnormal expression of phosphatidylserine on red blood cell (rbc) surface and consequent increased platelet activation and thrombin generation. In addition, a reduction of anticoagulants i.e. proteins C and S and antithrombin (AT) was demonstrated. However, coagulable state in patients with β-thalassemia following stem cell transplantation (SCT) has not been characterized.

DETAILED DESCRIPTION:
Hypercoagulable state is well recognized in patients with β-thalassemia. Evidences of hypercoagulability include abnormal expression of phosphatidylserine on red blood cell (rbc) surface and consequent increased platelet activation and thrombin generation. In addition, a reduction of anticoagulants i.e. proteins C and S and antithrombin (AT) was demonstrated. However, coagulable state in patients with β-thalassemia following stem cell transplantation (SCT) has not been characterized.Therefore, the objective is to compare coagulation markers and anticoagulants among β-thalassemics with and without SCT and normal control (NC).The subjects will be classified into 3 groups; β-thalassemia post SCT (Thal-SCT), β-thalassemia treated with regular transfusion (Thal-RT) and NC. Blood samples will be tested for annexin V (an index of abnormal expression of phosphatidylserine on rbc surface), markers of activation of coagulation system (thrombin antithrombin complex (TAT), prothrombin fragment (F1+2), and D-dimer) and anticoagulants (proteins C and S and AT).

ELIGIBILITY:
Inclusion Criteria:

Group 1: beta thalassemia major or beta thalassemia / Hb E who receive regular transfusion therapy (Thal- RT). The baseline Hct was more than 24% for at least 6 months.

Group 2: beta thalassemia major or beta thalassemia / Hb E post SCT (Thal-SCT) who were discontinued immunosuppressive drugs.

Group 3: Normal children (NC) who had normal Hb/Hct and MCV for age

Exclusion Criteria:

Children with beta thalassemia major or beta thalassemia / Hb E who have co-diseases such as immune hemolytic anemia, infection, or inflammatory diseases

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The subjects were classified into 3 groups; β-thalassemia post SCT (Thal-SCT), β-thalassemia treated with regular transfusion (Thal-RT) and NC.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Level of protein C,S and AT, TAT, P1+2 and D-dimer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nongnuch Sirachainan, MD, Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Department of Pediatrics, Ramathibodi hospital, Bangkok, Thailand